CLINICAL TRIAL: NCT02094417
Title: A Phase 2, Randomized, Open-Label, Parallel, Comparative, Dose-Finding Study to Evaluate the Efficacy and Safety of AMG531 in Aplastic Anemia Subjects With Thrombocytopenia Refractory to Immunosuppressive Therapy
Brief Title: A Phase 2 Study to Evaluate the Efficacy and Safety of AMG531 in Aplastic Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 531-KR001
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Results first posted 2021-02-15 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Aplastic Anemia
Keywords: Anemia, Aplastic; Thrombopoietin; Thrombocytopenia
MeSH Terms: conditions — Anemia, Aplastic; Jacobs syndrome; Thrombocytopenia | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- AMG531 (Dose 1) (Experimental)
  Interventions: Drug: AMG531
- AMG531 (Dose 2) (Experimental)
  Interventions: Drug: AMG531
- AMG531 (Dose 3) (Experimental)
  Interventions: Drug: AMG531
- AMG531 (Dose 4) (Experimental)
  Interventions: Drug: AMG531

INTERVENTIONS:
Drug: AMG531 — Subcutaneous, weekly injection

SUMMARY:
The present study will be conducted to evaluate the efficacy and safety of AMG531 and to determine the recommended initial dose of AMG531 on the basis of its efficacy and safety when it is administered subcutaneously (SC) to the Aplastic Anemia (AA) patients with immunosuppressive-therapy refractory thrombocytopenia and also to assess the pharmacokinetics of this product. Its efficacy and safety during the extension period beyond one year will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is diagnosed as AA and refractory to immunosuppressive therapy
* Platelet ≤ 30,000/μL

Exclusion Criteria:

* Concurrent active infection not adequately responding to appropriate therapy
* HIV positivity
* Bone marrow reticulin grade of > 1
* Clinically significant cardiac disease
* Arterial or venous thrombosis within the last 1 year before enrollment
* Other cause of thrombocytopenia
* AA with hemolytic predominant paroxysmal nocturnal hemoglobinuria (PNH)
* Uncontrolled diabetes
* Receiving any agent used to treat AA, including antithymocyte globulin (ATG) or ATG + cyclosporine within 6 months before starting study treatment and/or cyclosporine or anabolic hormone within 6 weeks before starting the study treatment
* History of PEG-rHuMGDF, recombinant human thrombopoietin, AMG531, and other thrombopoietin (TPO)-receptor agonist
* Who plans to conduct hematopoietic stem cell transplantation within 1 year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Korea, Republic of, Seoul, South Korea

REFERENCES:
- [Derived] Jang JH, Mitani K, Tomiyama Y, Miyazaki K, Nagafuji K, Usuki K, Uoshima N, Fujisaki T, Kosugi H, Matsumura I, Sasaki K, Kizaki M, Sawa M, Hidaka M, Kobayashi N, Ichikawa S, Yonemura Y, Murotani K, Shimizu M, Matsuda A, Ozawa K, Nakao S, Lee JW. Predictive factors of romiplostim response in patients with refractory aplastic anemia: data from two clinical trials. Ann Hematol. 2025 Aug;104(8):4003-4011. doi: 10.1007/s00277-025-06337-7. Epub 2025 Jul 1. PMID 40593138
- [Derived] Lee JW, Lee SE, Jung CW, Park S, Keta H, Park SK, Kim JA, Oh IH, Jang JH. Romiplostim in patients with refractory aplastic anaemia previously treated with immunosuppressive therapy: a dose-finding and long-term treatment phase 2 trial. Lancet Haematol. 2019 Nov;6(11):e562-e572. doi: 10.1016/S2352-3026(19)30153-X. Epub 2019 Aug 29. PMID 31474546

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 14 April 2014 through 28 November 2014 from two clinical centers (Seoul St. Mary's Hospital and Samsung Medical Center, Seoul, South Korea).
Groups:
- AMG531 (Dose 1): AMG531: 1 μg/kg, subcutaneous, once weekly
- AMG531 (Dose 2): AMG531: 3 μg/kg, subcutaneous, once weekly
- AMG531 (Dose 3): AMG531: 6 μg/kg, subcutaneous, once weekly
- AMG531 (Dose 4): AMG531: 10 μg/kg, subcutaneous, once weekly
Period: Overall Study
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 2) | AMG531 (Dose 3) | AMG531 (Dose 4)
Started | 7 | 9 | 9 | 10
Completed | 2 | 1 | 4 | 3
Not Completed | 5 | 8 | 5 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Eligibility criteria | 0 | 1 | 0 | 0
Not completed — No responder | 4 | 4 | 4 | 3
Not completed — Unable to conduct observations or assess | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- AMG531 (Dose 3): AMG531: 3 μg/kg, subcutaneous, once weekly
- AMG531 (Dose 2): AMG531: 6 μg/kg, subcutaneous, once weekly
- Total: Total of all reporting groups
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 3) | AMG531 (Dose 2) | AMG531 (Dose 4) | Total
Number analyzed (Participants) | 7 | 9 | 9 | 10 | 35
Age, Continuous [Median (Full Range); unit: years] | 45.0 [32 to 62] | 51.0 [33 to 60] | 50.0 [28 to 68] | 51.5 [33 to 76] | 49.0 [28 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 4 | 6 | 18
  Male | 5 | 3 | 5 | 4 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline platelet count [Mean (Standard Deviation); unit: cells 10^9/L] | 7.5 (3.6) | 9.9 (8.5) | 10.7 (6.9) | 9.8 (5.1) | 9.6 (6.2)
Baseline hemoglobin concentration [Mean (Standard Deviation); unit: g/dL] — Population: There was no data.
  g/dL
    number analyzed (Participants) | 4 | 7 | 4 | 6 | 21
    (all) | 6.73 (0.57) | 6.63 (0.71) | 5.95 (1.04) | 6.50 (2.14) | 6.48 (1.26)
Baseline neutrophil count [Mean (Standard Deviation); unit: cells 10^9/L] | 0.8902 (0.3606) | 0.9611 (0.6784) | 0.8756 (0.5000) | 0.9215 (0.3836) | 0.9136 (0.4797)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving a Platelet Response at Week 9
Description: The proportion of subjects achieving a platelet response at Week 9, and two-sided 95% confidence interval will be calculated. Platelet response is defined as 1) achieving absolute platelet increase of ≥ 20x10^9/L above baseline or 2) increase to ≥ 10x10^9/L and by at least 100% from baseline.
Time Frame: At week 9
Population: All efficacy analyses were carried out using the Per Protocol Set, which was defined as all enrolled subjects who received ≥6 times of the specified dose, with no major violation in the initial dose evaluation period. The Overall Number of Participants Analyzed is not consistent with numbers provided in the Participant Flow module because the Participant Flow module has been recorded based on the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 2) | AMG531 (Dose 3) | AMG531 (Dose 4)
Number analyzed (Participants) | 7 | 7 | 9 | 10
Participants | 0 | 0 | 3 | 7

2. Secondary Outcome: Proportion of Subjects Achieving a Platelet Response
Description: The proportion of subjects with a platelet response in any time during the initial dose evaluation period, Week 1 through Week 12, Week 1 through Week 16, Week 1 through Week 24, Week 1 through Week 52, Week 1 through Week 104 and Week 1 through Week 156.
Time Frame: Initial dose evaluation period (Week 9), Week 12, Week 16, Week 24, Week 52, Week 104, and Week 156
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 2) | AMG531 (Dose 3) | AMG531 (Dose 4)
Number analyzed (Participants) | 7 | 7 | 9 | 10
Participants
  Initial dose evaluation period | 3 | 3 | 6 | 10
  Week 1 - Week 12 | 4 | 4 | 7 | 10
  Week 1 - Week 16 | 4 | 4 | 7 | 10
  Week 1 - Week 24 | 6 | 4 | 8 | 10
  Week 1 - Week 52 | 6 | 5 | 8 | 10
  Week 1 - Week 104 | 6 | 5 | 8 | 10
  Week 1 - Week 156 | 6 | 5 | 8 | 10

3. Secondary Outcome: Proportion of Subjects Achieving Platelet Transfusion Independency
Description: The proportion of subjects achieving platelet transfusion independency in any time during the initial dose evaluation period , Week 1 through Week 12, Week 1 through Week 16, Week 1 through Week 24, Week 1 through Week 52, Week 1 through Week 104, and Week1 through Week 156 will be calculated in the same manner as the primary variables (The number of subjects discontinued or subjects who have missing data will not be calculated). Platelet transfusion independence is defined as achieving transfusion free period of at least 8 consecutive weeks (56 days).
Time Frame: Initial dose evaluation period (Week 9), Week 12, Week 16, Week 24, Week 52, Week 104, and Week 156
Population: With respcet to platelet transfusion indendpendence, the proportion will be calculated based on all subjcets in each analysis set and all subjects receving platelet transfusion as a pretreatment 8 weeks prior to the first AMG531 administration respectively.
Measure: Count of Participants; unit: Participants
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 2) | AMG531 (Dose 3) | AMG531 (Dose 4)
Number analyzed (Participants) | 7 | 7 | 9 | 10
Participants
  All subjects : Initial dose evaluation period | 0 | 2 | 0 | 2
  All subjects : Week 1 - Week 12 | 0 | 2 | 1 | 4
  All subjects : Week 1 - Week 16 | 0 | 2 | 2 | 4
  All subjects : Week 1 - Week 24 | 1 | 2 | 3 | 6
  All subjects : Week 1 - Week 52 | 2 | 2 | 3 | 6
  All subjects : Week 1 - Week 104 | 2 | 2 | 3 | 6
  All subjects : Week 1 - Week 156 | 2 | 2 | 3 | 6
  Subjects with TF : Initial dose evaluation period: number analyzed (Participants) | 5 | 4 | 6 | 6
  Subjects with TF : Initial dose evaluation period | 0 | 2 | 0 | 2
  Subjects with TF : Week 1 - Week 12 | 0 | 2 | 1 | 4
  Subjects with TF : Week 1 - Week 16 | 0 | 2 | 2 | 4
  Subjects with TF : Week 1 - Week 24 | 1 | 2 | 3 | 6
  Subjects with TF : Week 1 - Week 52 | 2 | 2 | 3 | 6
  Subjects with TF : Week 1 - Week 104 | 2 | 2 | 3 | 6
  Subjects with TF : Week 1 - Week 156 | 2 | 2 | 3 | 6

4. Secondary Outcome: Proportion of Subjects Achieving Erythroid Response and/or Neutrophil Response
Description: The proportion of subjects with erythroid response, neutrophil response and erythroid and/or neutrophil response in any time during the initial dose evaluation period, Week 1 through Week 12, Week 1 through Week 16, Week 1 through Week 24, Week 1 through Week 52, Week 1 through Week 104, and Week1 through Week 156 will be calculated in the same manner as the primary variables (The number of subjects discontinued or subjects who have missing data will not be calculated).
Time Frame: Initial dose evaluation period (Week 9), Week 12, Week 16, Week 24, Week 52, Week 104, and Week 156
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 2) | AMG531 (Dose 3) | AMG531 (Dose 4)
Number analyzed (Participants) | 7 | 7 | 9 | 10
Participants
  Erythroid Response : Initial dose evaluation period | 0 | 2 | 1 | 3
  Erythroid Response : Week 1 - Week 12 | 0 | 4 | 4 | 4
  Erythroid Response : Week 1 - Week 16 | 3 | 4 | 4 | 4
  Erythroid Response : Week 1 - Week 24 | 5 | 5 | 7 | 5
  Erythroid Response : Week 1 - Week 52 | 6 | 5 | 7 | 7
  Erythroid Response : Week 1 - Week 104 | 6 | 5 | 7 | 7
  Erythroid Response : Week 1 - Week 156 | 6 | 5 | 7 | 7
  Neutrophil Response : Initial dose evaluation period | 1 | 3 | 4 | 6
  Neutrophil Response : Week 1 - Week 12 | 1 | 3 | 5 | 6
  Neutrophil Response : Week 1 - Week 16 | 2 | 4 | 5 | 6
  Neutrophil Response : Week 1 - Week 24 | 4 | 4 | 5 | 7
  Neutrophil Response : Week 1 - Week 52 | 4 | 5 | 5 | 7
  Neutrophil Response : Week 1 - Week 104 | 4 | 5 | 5 | 7
  Neutrophil Response : Week 1 - Week 156 | 4 | 5 | 5 | 7
  Erythroid response and/or Neutrophil response : Initial dose evaluation period | 1 | 4 | 5 | 7
  Erythroid response and/or Neutrophil response : Week 1 - Week 12 | 1 | 5 | 7 | 7
  Erythroid response and/or Neutrophil response : Week 1 - Week 16 | 4 | 5 | 7 | 7
  Erythroid response and/or Neutrophil response : Week 1 - Week 24 | 7 | 6 | 8 | 8
  Erythroid response and/or Neutrophil response : Week 1 - Week 52 | 7 | 6 | 8 | 8
  Erythroid response and/or Neutrophil response : Week 1 - Week 104 | 7 | 6 | 8 | 8
  Erythroid response and/or Neutrophil response : Week 1 - Week 156 | 7 | 6 | 8 | 8

5. Secondary Outcome: Duration of Platelet Response and Time to Platelet Response
Description: For subjects with a platelet response in any time, time to the initial platelet response and duration of platelet response will be summarized Time to the initial platelet response will be calculated as sampling date (response achieved) minus first dose date of study drug plus 1.
  Duration of platelet response will be calculated as the maximum of the duration of platelet response for each subject, each duration of response calculated as the date when response is disappeared minus the date when response is achieved. The censoring date is defined as the date of the last Platelet examination or EOS whichever archives first.
Time Frame: Initial dose evaluation period (Week 9), Week 12, Week 16, Week 24, Week 52, Week 104, and Week 156
Population: A total of 29 subjects achieved a platelet response and the median duration of the platelet response was 77.0 days (range: 5 to 959 days). For the 29 subjects who achieved a platelet response, the median time to the initial platelet response was 43 days (range: 8 to 219 days).
Measure: Median (Full Range); unit: days
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 2) | AMG531 (Dose 3) | AMG531 (Dose 4)
Number analyzed (Participants) | 7 | 7 | 9 | 10
days
  Duration of platelet response: number analyzed (Participants) | 6 | 5 | 8 | 10
  Duration of platelet response | 24.5 [14 to 506] | 21.0 [9 to 862] | 503.5 [7 to 959] | 131.0 [5 to 886]
  Time to the initial platelet response: number analyzed (Participants) | 6 | 5 | 8 | 10
  Time to the initial platelet response | 59.0 [8 to 127] | 44.0 [15 to 219] | 53.5 [22 to 134] | 41.0 [36 to 50]

6. Secondary Outcome: Proportion of Subjects Achieving Tri-lineage Responses
Description: Tri-lineage response is defined in those achieving platelet response, erythroid response, and neutrophil response all together. The proportion of subjects with tri-lineage response will be calculated in the same manner as the primary variables. Time to tri-lineage response will be summarized in the same manner as time to platelet response. Time to tri-lineage response is defined as duration of the time from Day 1 to the date of platelet response, erythroid response or neutrophil response whichever achieves last in Visit.
Time Frame: Initial dose evaluation period (Week 9), Week 12, Week 16, Week 24, Week 52, Week 104, and Week 157
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 2) | AMG531 (Dose 3) | AMG531 (Dose 4)
Number analyzed (Participants) | 7 | 7 | 9 | 10
Participants
  Week 9 | 0 | 0 | 0 | 0
  Week 13 | 0 | 0 | 0 | 0
  Week 17 | 0 | 1 | 0 | 0
  Week 25 | 1 | 1 | 1 | 1
  Week 27 | 0 | 1 | 2 | 0
  Week 53 | 1 | 1 | 2 | 1
  Week 105 | 1 | 1 | 2 | 1
  Week 157 | 1 | 1 | 3 | 0

7. Secondary Outcome: Duration of Study Drug Discontinuation While Maintaining Stable Response
Description: The longest duration of study drug discontinuation in subjects while maintaining a stable response is summarized
Time Frame: Initial dose evaluation period (Week 9), Week 12, Week 16, Week 24, Week 52, Week 104, and Week 156
Population: 3/33 (9.1%) subjects (who maintained blood cell response) discontinued the study drug during Week 1 to Week 156.
Measure: Median (Full Range); unit: days
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 2) | AMG531 (Dose 3) | AMG531 (Dose 4)
Number analyzed (Participants) | 0 | 0 | 2 | 1
days |  |  | 273.0 [56 to 490] | 483.0 [483 to 483]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: This section focuses primarily on treatment-emergent AEs (TEAEs), defined as any untoward medical occurrence in subjects who received AMG531. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom or disease, regardless of causal relationship to AMG531.
Arm/Group | AMG531 (Dose 1) | AMG531 (Dose 2) | AMG531 (Dose 3) | AMG531 (Dose 4)
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/9 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/7 | 2/9 | 2/9 | 3/10
Other Adverse Events (participants affected / at risk) | 3/7 | 5/9 | 7/9 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMG531 (Dose 1) (N=7) | AMG531 (Dose 2) (N=9) | AMG531 (Dose 3) (N=9) | AMG531 (Dose 4) (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMG531 (Dose 1) (N=7) | AMG531 (Dose 2) (N=9) | AMG531 (Dose 3) (N=9) | AMG531 (Dose 4) (N=10)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin conjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT02094417/Prot_SAP_000.pdf